CLINICAL TRIAL: NCT04817007
Title: A Phase 1b/2 Study of BMS-986158 Monotherapy and in Combination With Either Ruxolitinib or Fedratinib in Participants With DIPSS-Intermediate or High Risk Myelofibrosis
Brief Title: A Study to Assess the Safety and Tolerability of BMS-986158 Alone and in Combination With Either Ruxolitinib or Fedratinib in Participants With Blood Cancer (Myelofibrosis)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA011-023; 2020-002071-35 (EudraCT Number)
Expanded Access: NCT05301972 (No longer available)
Record Dates: First submitted 2021-03-18; First posted 2021-03-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis
Keywords: BMS-986158; Fedratinib; Myelofibrosis; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1A: BMS-986158 + Ruxolitinib (Experimental)
  Interventions: Drug: BMS-986158; Drug: Ruxolitinib
- Part 1B: BMS-986158 + Fedratinib (Experimental)
  Interventions: Drug: BMS-986158; Drug: Fedratinib
- Part 2A1: BMS-986158 + Ruxolitinib (Experimental)
  Interventions: Drug: BMS-986158; Drug: Ruxolitinib
- Part 2B1: BMS-986158 + Fedratinib (Experimental)
  Interventions: Drug: BMS-986158; Drug: Fedratinib
- Part 2B2: BMS-986158 Mono and/or (BMS-986158 + Fedratinib), if applicable (Experimental)
  Interventions: Drug: BMS-986158; Drug: Fedratinib
- Part 2A2 Add-On: BMS-986158 + Ruxolitinib (Experimental)
  Interventions: Drug: BMS-986158; Drug: Ruxolitinib
- Part 2A3: BMS-986158 + Ruxolitinib (Experimental)
  Interventions: Drug: BMS-986158; Drug: Ruxolitinib

INTERVENTIONS:
Drug: BMS-986158 — Specified dose on specified days
Drug: Ruxolitinib — Specified dose on specified days
  Other Names: Jakafi®
  Arms: Part 1A: BMS-986158 + Ruxolitinib; Part 2A1: BMS-986158 + Ruxolitinib; Part 2A2 Add-On: BMS-986158 + Ruxolitinib; Part 2A3: BMS-986158 + Ruxolitinib
Drug: Fedratinib — Specified dose on specified days
  Arms: Part 1B: BMS-986158 + Fedratinib; Part 2B1: BMS-986158 + Fedratinib; Part 2B2: BMS-986158 Mono and/or (BMS-986158 + Fedratinib), if applicable

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of BMS-986158 alone and in combination with either Ruxolitinib or Fedratinib in participants with Dynamic International Prognostic Scoring System (DIPSS)-intermediate or high risk blood cancer. Part 1 consists of BMS-986158 in combination with either Ruxolitinib or Fedratinib and Part 2 consists of BMS-986158 in combination with either Ruxolitinib or Fedratinib and BMS-986158 alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis (PMF), post-essential thrombocythemia (ET) or post-polycythemia vera (PV) myelofibrosis
* Treatment-related toxicities from prior therapy resolved to Grade 1 or pre-treatment baseline or determined to be irreversible prior to study treatment
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women who are pregnant or breastfeeding at screening
* Any significant acute or uncontrolled chronic medical illness

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 52 months
Incidence of serious adverse events (SAEs) | Up to 52 months
Incidence of AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria | Up to 26 months
Incidence of AEs leading to discontinuation | Up to 52 months
Incidence of death | Up to 52 months

SECONDARY OUTCOMES:
Spleen volume reduction (SVR) at end of Cycle 6 assessed by Blinded Independent Central Review (BICR) | Up to 175 days
Response rate defined as proportion of participants with SVR ≥ 35% by MRI (preferred) or CT (if MRI is contraindicated and if CT is allowed by local guidelines) assessed by BICR | Up to 175 days
SVR at end of Cycle 3 and 6 assessed by BICR | Up to 175 days
Response rate defined as proportion of participants with SVR ≥ 25% by MRI (preferred) or CT (if MRI is contraindicated and if CT is allowed by local guidelines) assessed by BICR | Up to 175 days
Symptom response rate (SRR) based on total symptom score (TSS) measured by Myelofibrosis Symptom Assessment Form (MFSAF) | Up to 175 days
Additional measures based on TSS measured by MFSAF | Up to 175 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (8):
  - Local Institution - 0069, Newport Beach, California
  - Local Institution - 0090, Lake Mary, Florida
  - Local Institution - 0043, New Orleans, Louisiana
  - Local Institution - 0038, Worcester, Massachusetts
  - Local Institution - 0033, Ann Arbor, Michigan
  - Local Institution - 0045, Hackensack, New Jersey
  - Local Institution - 0076, Chapel Hill, North Carolina
  - Local Institution - 0042, Pittsburgh, Pennsylvania
- Australia (6):
  - Local Institution - 0036, Blacktown, New South Wales
  - Local Institution - 0032, Wollongong, New South Wales
  - Local Institution - 0007, East Melbourne, Victoria
  - Local Institution - 0006, Heidelberg, Victoria
  - Local Institution - 0041, Nedlands, Western Australia
  - Local Institution - 0015, West Perth, Western Australia
- France (5):
  - Local Institution - 0030, Brest
  - Local Institution - 0008, Marseille
  - Local Institution - 0027, Nice
  - Local Institution - 0011, Paris
  - Local Institution - 0010, Villejuif
- Germany (5):
  - Local Institution - 0068, Erding, Bavaria
  - Local Institution - 0039, Essen, North Rhine-Westphalia
  - Local Institution - 0040, Chemnitz, Saxony
  - Local Institution - 0035, Halle, Saxony-Anhalt
  - Local Institution - 0050, Lübeck, Schleswig-Holstein
- Greece (2):
  - Local Institution - 0061, Chaïdári, Attikí
  - Local Institution - 0047, Thessaloniki, Thessaloníki
- Hungary (4):
  - Local Institution - 0073, Szeged, Csongrád megye
  - Local Institution - 0072, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Local Institution - 0075, Budapest
  - Local Institution - 0074, Debrecen
- Israel (5):
  - Local Institution - 0086, Beersheba, Southern District
  - Local Institution - 0016, Jerusalem
  - Local Institution - 0018, Petah Tikva
  - Local Institution - 0017, Ramat Gan
  - Local Institution - 0019, Tel Aviv
- Italy (4):
  - Local Institution - 0003, Bologna
  - Local Institution - 0002, Brescia
  - Local Institution - 0001, Florence
  - Local Institution - 0012, Verona
- Poland (2):
  - Local Institution - 0077, Słupsk, Pomeranian Voivodeship
  - Local Institution - 0062, Gdansk
- Romania (3):
  - Local Institution - 0052, Bucuresti, Cluj
  - Local Institution - 0083, Bucharest
  - Local Institution - 0051, Cluj-Napoca
- South Korea (3):
  - Local Institution - 0049, Seongnam, Kyǒnggi-do
  - Local Institution - 0048, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0053, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (6):
  - Local Institution - 0020, Badalona, Barcelona [Barcelona]
  - Local Institution - 0029, Santander, Cantabria
  - Local Institution - 0054, Madrid, Madrid, Comunidad de
  - Local Institution - 0026, Madrid
  - Local Institution - 0021, Salamanca
  - Local Institution - 0094, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04817007.html